CLINICAL TRIAL: NCT01336101
Title: Evaluation of Efficacy of the EPIC™ Self-Expanding Nitinol Vascular Stent With Delivery System -The SUMMIT Registry
Brief Title: Evaluation of Efficacy of the EPIC™ Self-Expanding Nitinol Vascular Stent
Acronym: SUMMIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Provascular GmbH (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prov 01 - 2011; ISROTH10001 (Other Grant/Funding Number: Boston Scientific); U1111-1121-6816 (Registry Identifier: Universal Trial Number)
Record Dates: First submitted 2011-04-12; First posted 2011-04-15 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Peripheral Arterial Diseases; Superficial Femoral Artery Stenosis
Keywords: PAD; SFA
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SFA stenting (Other)
  Interventions: Device: EPIC™ Self-Expanding Nitinol Vascular Stent

INTERVENTIONS:
Device: EPIC™ Self-Expanding Nitinol Vascular Stent — SFA/Popliteal Artery stenting

SUMMARY:
The intent of this clinical registry is to demonstrate the efficacy of the EPIC™ stent in patients with superficial femoral/ popliteal artery disease.

100 patients with symptomatic femoropopliteal artery lesion will be enrolled in the study and shall undergo 4 visits during the trial -a pre-procedure visit, procedure visit at which time the stent will be placed, and follow-up visits at 6 and 12 months.

Study hypothesis: The EPIC™ Self-Expanding Nitinol Vascular Stent with Delivery System will be efficacious in patients with Superficial Femoro/Popliteal Artery disease.

DETAILED DESCRIPTION:
The SUMMIT Registry addresses the treatment of peripheral arterial disease (PAD).

PAD represents a major challenge to physicians in treating the Superficial Femoral (SFA) and Popliteal arteries. These vessels are exposed to enormous mechanical stress what represents a harsh environment for any endovascular device. During flexing of the knee, the SFA/Popliteal arteries can bend, rotate, elongate and compress dramatically. An ideal stent designed for use in the SFA/Popliteal arteries would offer great ranges of movement while adequately supporting the arteries.

Subject of study is the EPIC™ Femoropopliteal Self-Expanding Stent System which provides a great range of motions for a highly flexible femoral artery while adequately supporting the vessel.

Primary objective is to evaluate the efficacy of the device in treating lesions of the SFA/Popliteal artery.

The project is a multi-centre open label study. Primary efficacy parameter will be assessed by measuring the in-stent binary stenosis using duplex ultrasound at 6 and 12 months after the stent placement. Binary restenosis is defined as a peak systolic velocity ratio (PSVR) ≥2.5:1.

Anticipated study duration is 18 months: 6 months recruiting and 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, male or female, must be between the ages of 18 to 85 years inclusive at the time of consent. A female of childbearing potential may be enrolled, provided she has a negative pregnancy test at Screening.
* Subjects must give written informed consent prior to participation in the study and must understand the purpose of this study and be willing to adhere to the study procedures described in this protocol.
* Rutherford Classification Category 2-4
* Single de novo lesion in the superficial femoro/popliteal artery
* Disease segment length ≤150mm
* >70% diameter stenosis and occlusion
* Patent ipsilateral iliac artery
* Patent ipsilateral popliteal artery and at least 1 patent tibial artery in continuity to ankle
* Target reference vessel diameter 3.5-7.5 mm

Exclusion Criteria:

* Target lesion previously treated with a stent or surgery.
* Rutherford Classification Category 0, 1, 5 or 6.
* Inability to tolerate antithrombotic or antiplatelet therapies.
* Pregnancy.
* Other co morbidity risks which in the opinion of the investigator limit longevity or likelihood of complying with protocol follow up.
* Serum creatinine > 2.5 mg/dL.
* Myocardial infarction or stroke within 90 days of enrollment.
* Hypercoagulable state.
* Uncontrollable hypertension.
* Patients currently enrolled in any other clinical trial(s).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-04; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
efficacy of the EPIC™ Stent as measured by the in-stent binary restenosis using duplex ultrasound (DUS) | at 6 months after procedure
  Binary restenosis is defined as a peak systolic velocity ratio (PSVR) ≥2.5:1.
efficacy of the EPIC™ Stent as measured by the in-stent binary restenosis using duplex ultrasound (DUS) | at 12 months after procedure
  Binary restenosis is defined as a peak systolic velocity ratio (PSVR) ≥2.5:1.

SECONDARY OUTCOMES:
Technical Success | after stent placement intra-procedural via angiographic images (day 1)
  defined as the ability to implant the stent with a residual angiographic stenosis no greater than 30%.

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, Principal Investigator — Park-Krankenhaus Leipzig
Locations (4):
- Germany (4):
  - Herz-Zentrum, Bad Krozingen
  - Weisseritztal-Kliniken, Freital
  - Park-Krankenhaus, Leipzig
  - Medinos Kliniken, Sonneberg

REFERENCES:
- [Derived] Werner M, Piorkowski M, Thieme M, Nanning T, Beschorner U, Rastan A, Zeller T, Scheinert D. SUMMIT registry: one-year outcomes after implantation of the EPIC self-expanding nitinol stent in the femoropopliteal segment. J Endovasc Ther. 2013 Dec;20(6):759-66. doi: 10.1583/13-4430R.1. PMID 24325691